CLINICAL TRIAL: NCT01934101
Title: A Phase 1 Double-blind, Randomised, Placebo-controlled, Dose Escalating Study to Assess the Safety and Tolerability of Single and Multiple Oral Doses of CHR-5154 and the Effect of the Fasted and Fed State on Pharmacokinetics of CHR-5154 and CHR-5426 in Healthy Male Volunteers
Brief Title: Phase 1 Dose Escalating Study to Assess Safety, Tolerability, Food Effect and PK of CHR-5154 in Healthy Male Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Following the emergence of an unexpected pharmacodynamic effect, the sponsor has decided to conclude the study early without fully achieving its objective
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201302
Record Dates: First submitted 2013-07-15; First posted 2013-09-04 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CHR-5154 (Experimental): CHR-5154
  Interventions: Drug: CHR-5154
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CHR-5154 — CHR-5154
  Arms: CHR-5154
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Primary Objective:

• To determine the safety and tolerability of single and multiple ascending oral doses of CHR-5154 in healthy volunteers.

Secondary Objectives:

* To determine the pharmacokinetic profile of CHR-5154 and its metabolite CHR-5426.
* To compare the pharmacokinetic profile of CHR-5154 and CHR-5426 after a single dose of CHR-5154 in the fed and fasted state.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteers aged 18-45.
2. Non-smokers from at least three months before receiving the first dose of study drug and for the duration of the study.
3. Body mass index (BMI) ≥ 18 and ≤ 32 kg/m2.
4. Body weight ≥ 50 kg and ≤ 120 kg at screening.
5. Able to voluntarily provide written informed consent to participate in the study.
6. Must understand the purposes and risks of the study and agree to follow the restrictions and schedule of procedures as defined in the protocol, as confirmed during the informed consent process.
7. Sexually active male volunteers must use two highly effective methods of contraception with their partners throughout the study and for 90 days after completion of the study.
8. Male volunteers must not donate sperm during the study and for 90 days after completion of the study.
9. Must be willing to consent to have data entered into The Over Volunteering Prevention System (TOPS).
10. The volunteer's primary care physician must confirm that there is nothing in their medical history that would preclude their enrolment into this clinical study

Exclusion Criteria:

1. Volunteers with history or presence of significant cardiovascular disease, pulmonary, hepatic, gallbladder or biliary tract, renal, haematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, psychiatric disease or current infection.
2. Laboratory values at screening or baseline which are deemed to be clinically significant.
3. QTcF greater than 450 msec at screening.
4. Positive for human immunodeficiency virus (HIV), hepatitis B or hepatitis C.
5. Current or history of drug or alcohol abuse or a positive drugs of abuse or alcohol test at screening or check-in.
6. Participation in a clinical drug study during the 90 days preceding the initial dose in this study.
7. Any clinically significant illness within 30 days prior to study drug administration.
8. Donation of blood or blood products within 90 days prior to study drug administration, or at any time during the study, except as required by this protocol.
9. Volunteers who have a history or presence of any significant drug allergy.
10. Use of any prescription or over-the-counter medication (including vitamins, herbal and mineral supplements) within 30 days prior to study drug administration until the end of the study, with the exception of occasional paracetamol approved by the Investigator.
11. Strenuous exercise, as judged by the Investigator, within 72 hours prior to screening, within 72 hours prior to study drug administration and for the duration of the study until after the post-study medical.
12. Weekly alcohol intake exceeding the equivalent of 21 units per week.
13. Consumption of alcoholic beverages within 24 hours prior to study drug administration and during study confinement.
14. Consumption of caffeine or xanthine-containing products within 24 hours prior to confinement and during study confinement.
15. Consumption of grapefruit, grapefruit juice, Seville oranges, Seville orange marmalade or other products containing grapefruit or Seville oranges within 7 days prior to confinement and during study confinement.
16. Volunteers who, in the opinion of the Investigator, are unsuitable for participation in the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2013-08-12 (Actual); Primary Completion 2014-05-28 (Actual); Study Completion 2014-05-28 (Actual)

PRIMARY OUTCOMES:
Number of volunteers with adverse events | upto 10 days in Single ascending dose phase and 16 days in the Multiple ascending dose phase

SECONDARY OUTCOMES:
To determine the pharmacokinetic profile of CHR-5154 and its metabolite CHR-5426. | upto 48 hrs post dose
To compare the pharmacokinetic profile of CHR-5154 and CHR-5426 after a single dose of CHR-5154 in the fed and fasted state. | Upto 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Belfast, United Kingdom

REFERENCES:
- See also: Results for study 201302 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/201302?search=study&study_ids=201302#rs